CLINICAL TRIAL: NCT05317468
Title: Pilot Randomized Controlled Trial to Assess Satisfaction With Contraceptive Counseling Using Telephone Versus Video Telehealth Visits
Brief Title: Assessing Satisfaction With Contraceptive Counseling Using Telephone Versus Video Telehealth Visits
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Washington University School of Medicine (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: 202203067
Record Dates: First submitted 2022-03-23; First posted 2022-04-07 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Contraception; Health Care Utilization
MeSH Terms: conditions — Patient Acceptance of Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Video (Experimental): Patients will complete contraceptive counseling using a video-based platform. Patients and counselors will have an audio and video connection.
  Interventions: Other: Contraceptive Counseling
- Telephone (Experimental): Patients will complete contraceptive counseling on a telephone call. Patients and counselors will have an audio connection only.
  Interventions: Other: Contraceptive Counseling

INTERVENTIONS:
Other: Contraceptive Counseling — Patients will receive contraceptive counseling to review all available contraceptive methods prior to their visit with a clinician.

SUMMARY:
The Contraceptive Choice Center (C3) will compare the patient experience between patients receiving contraceptive counseling using a telephone versus video telehealth model.

DETAILED DESCRIPTION:
The Contraceptive Choice Center (C3) will offer contraceptive counseling to patients via telehealth. Participants will be randomized to receive counseling via video or telephone. We will compare patient satisfaction with contraceptive counseling, receipt of desired contraceptive method, and identification of barriers with technology use.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and read English
* Access to video-capable technology

Exclusion Criteria:

* Incarceration
* Unable to provide informed consent secondary to language barrier or cognitive limitation

Min Age: 14 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 214 (Actual)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-14 (Actual); Study Completion 2023-06-26 (Actual)

PRIMARY OUTCOMES:
Patient Satisfaction Assessed by IQFP | Baseline
  Interpersonal Quality in Family Planning (IQFP) scale
  Continuous score: 11-55, higher scores indicate higher patient satisfaction Dichotomous: highest score (55) versus lower scores, highest score indicates highest patient satisfaction

SECONDARY OUTCOMES:
% of Patients Receiving Desired Contraceptive Method Assessed by Medical Record Review | 30 Days Post Baseline
% of Patients Reporting Barriers to Technology Use Assessed by Baseline Questionnaire | Baseline
  Percentage of patients reporting limited access to mobile telephone or computer with video capabilities, unreliable telephone or internet service, and environmental distractors (i.e. loud noises, lack of privacy)

CONTACTS AND LOCATIONS:
Overall Officials: Jennifer A Reeves, MD, MPH, Principal Investigator — Washington University School of Medicine
Locations (1):
- Washington University School of Medicine, St Louis, Missouri, United States

IPD SHARING:
Plan to Share IPD: No